CLINICAL TRIAL: NCT00586690
Title: Safety Trial of Natural Killer (NK) Cell Donor Lymphocyte Infusions(DLI) From 6/6 Human Leukocyte Antigen (HLA) Matched Family Member Following Nonmyeloablative Allogeneic Stem Cell Transplantation (ASCT)
Brief Title: Safety Trial of NK DLI From 6/6 HLA Matched Family Member Following Nonmyeloablative ASCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005124
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma
Keywords: Stem cell transplant; matched donor; NK infusion
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NK Cell Infusion (Experimental): Natural Killer (NK) Cell infusion using CD56 monoclonal antibody
  Interventions: Device: NK Cell infusion using CD56 monoclonal antibody
- Donor Apheresis (Other): Apheresis repeated daily up to 3 days until target dose of cells reached (preferably without donor receiving growth factors). Cells were transfused immediately after collection and processing. If collections occurred during initial mobilization at the time of stem cell transplant, the donor was off growth factor for >24 hours. These extra cell collections from the donor were sufficient for the natural killer cells used in the trial. The cells were NK selected using a CD56 antibody (CliniMACS CD56 Reagent), CliniMACSplus instrument and CliniMACS tubing set provided by Miltenyi Biotec using the company protocol (Miltenyi Biotec Inc, Auburn, California). Pre and post processing cell count, viability, Hematopoietic Progenitor Cell Assay (HPCA) and flow analysis were done.
  Interventions: Procedure: Donor Apheresis

INTERVENTIONS:
Device: NK Cell infusion using CD56 monoclonal antibody — The cells from leukapheresis will be natural killer (NK) cell selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II acute graft versus host disease (aGVHD) at the time of infusion. Patients will be evaluated for toxicity and response until 20 weeks after the last NK Infusion.
  Other Names: CD56 monoclonal antibody
  Arms: NK Cell Infusion
Procedure: Donor Apheresis — Apheresis repeated daily up to 3 days until target dose of cells reached (preferably without donor receiving growth factors). Cells were transfused immediately after collection and processing. If collections occurred during initial mobilization at the time of stem cell transplant, the donor was off growth factor for >24 hours. These extra cell collections from the donor were sufficient for the natural killer cells used in the trial. The cells were NK selected using a CD56 antibody (CliniMACS CD56 Reagent), CliniMACSplus instrument and CliniMACS tubing set provided by Miltenyi Biotec using the company protocol (Miltenyi Biotec Inc, Auburn, California). Pre and post processing cell count, viability, Hematopoietic Progenitor Cell Assay (HPCA) and flow analysis were done.
  Arms: Donor Apheresis

SUMMARY:
Evaluate the safety of natural killer (NK) cell infusion using CD56 monoclonal antibody selected with Miltenyi Biotec system following nonmyeloablative stem cell transplantation (SCT) from matched donors. This pilot study will evaluate toxicity including mortality, occurrence of acute graft versus host disease and other severe toxicity.

DETAILED DESCRIPTION:
The use of non-selected donor lymphocyte infusions (DLIs) (to help early immune recovery and induce antitumor response) following nonmyeloablative allogeneic stem cell transplantation (ASCT) is also complicated by the risk of acute graft versus host disease (aGVHD) with 30-40% of patients experiencing grade III-IV aGVHD. Data suggests that the use of natural killer (NK) cells (instead of nonselected DLIs) in this setting may mediate a graft versus tumor (GVT) effect independently of aGVHD.

This pilot study is designed to evaluate the efficacy and toxicity of donor natural killer (NK) cell selection and infusion following nonmyeloablative allogeneic stem cell transplantation (ASCT) from matched donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with who have undergone a non-myeloablative allogeneic transplant, using a 6/6 human leukocyte antigen (HLA) matched sibling donor. Measureable disease is not needed at study entry.
* Performance status must be Karnofsky 50-100%.
* Donor cellular engraftment of at least 2.5% from the non-myeloablative procedure.
* ≤ Grade 2 acute Graft versus Host Disease (aGvHD) at time of infusion of natural killer (NK) cell infusion. Patients with treated aGVHD must be on a stable dose of therapy (no increase in immunosuppressive therapy for the 2 weeks before planned natural killer cell infusion [NKI]). The dosage/level of immunosuppressive therapy at the time of NKI should be no greater than 1 mg/kg of prednisone daily or mycophenolate 1000 mg bid daily or cyclosporine with a target level of 200 or equivalent.
* Estimated survival at least 8 weeks.
* Age > or equal to 18 years of age.

Exclusion Criteria:

* Pregnant or lactating women,
* Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance to this protocol.
* Patients who had biopsy proven overall Grade 4 GVHD lasting longer than 7 days, from the non-myeloablative therapy, are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-05; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Result] Rizzieri DA, Storms R, Chen DF, Long G, Yang Y, Nikcevich DA, Gasparetto C, Horwitz M, Chute J, Sullivan K, Hennig T, Misra D, Apple C, Baker M, Morris A, Green PG, Hasselblad V, Chao NJ. Natural killer cell-enriched donor lymphocyte infusions from A 3-6/6 HLA matched family member following nonmyeloablative allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2010 Aug;16(8):1107-14. doi: 10.1016/j.bbmt.2010.02.018. Epub 2010 Feb 24. PMID 20188202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty five participants were recruited through the Adult Bone Marrow Transplant Program at Duke University Medical Center. Recruitment began in May, 2005 and ended in April, 2010. Patients who met the eligibility criteria were approached about the study and informed consent was conducted for those who agreed.
Pre-assignment Details: Prior to initiating therapy, donors and subjects will have complete history, physical exam, routine laboratory tests, and/or radiographic tests. Recipients may have Bone marrow aspirate/biopsy repeated to check for prior abnormalities. If disease progression present, patient didn't continue with treatment.
Groups:
- Donor Apheresis: Leukapheresis was repeated daily up to 3 days until the target dose of cells was reached (preferably without donor receiving growth factors). When possible, cells were transfused immediately after collection and processing. If collections occurred during initial mobilization at the time of stem cell transplant, the donor was off growth factor for >24 hours. These collections, which are extra cells collected from the donor following initial collections for transplant were sufficient for the natural killer cells used in the trial. The cells were NK selected using a CD56 antibody (CliniMACS CD56 Reagent), CliniMACSplus instrument and CliniMACS tubing set provided by Miltenyi Biotec using the company protocol (Miltenyi Biotec Inc, Auburn, California). Pre and post processing cell count, viability, Hematopoietic Progenitor Cell Assay (HPCA) and flow analysis were done.
Period: Overall Study
Arm/Group | NK Cell Infusion | Donor Apheresis
Started | 21 (Four consented subjects were screen failures.) | 22
Completed | 5 | 22
Not Completed | 16 | 0
Not completed — Death | 2 | 0
Not completed — Disease Progression | 10 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lab can't accommodate | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible adult patients were those who engrafted following a fludarabine based T cell depleted non-myeloablative allogeneic transplant regimen with alemtuzumab. Donors were the same HLA 6/6 matched family member used for the allogeneic transplantation.
Groups:
- NK Cell Infusion: Natural Killer (NK) Cell infusion using CD56 monoclonal antibody: The cells from leukapheresis will be natural killer (NK) cell selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II acute graft versus host disease (aGVHD) at the time of infusion.
- Total: Total of all reporting groups
Arm/Group | NK Cell Infusion | Donor Apheresis | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 24 | 21 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 22 | 47
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Evaluate the toxicity post-infusion including mortality, occurrence of acute graft versus host disease (GVHD) and other severe toxicity until a minimum of 8 weeks following the last infusion, then at least monthly for 3 additional months. Unacceptable toxicity was defined as grade ≥ III aGVHD of the gut or liver or Grade 4 aGVHD of the skin lasting > 7 days; other Grade 4 toxicity from the procedure in the major organs that lasted > 5 days; or treatment-related mortality (TRM). Though these infusions are provided early following transplantation and severe toxicity could still have occurred due to the primary transplant procedure, for this study any aGVHD or other toxicities occurring after the first day of infusion of the natural killer (NK) cell enriched Donor Lymphocyte Infusions (DLIs) is considered here as study related.
Time Frame: 5 months
Population: Participants who completed cell infusion.
Measure: Number; unit: participants
Groups:
- NK Cell Infusion: Natural Killer (NK) Cell infusion using CD56 monoclonal antibody:
  The cells from leukapheresis will be NK cell selected using a CD56 antibody and a cell column system provided by Miltenyi Biotec. The target cell dose for each NK cell infusion will be up to 1 X 10(7) CD56+ cells/kg patient weight with less than 0.5 X 10(6) CD3+ cells/kg patient weight. The first NK cell infusion will be administered 6 weeks post transplant in patients who have ≤ grade II acute graft versus host disease (aGVHD) at the time of infusion.
Arm/Group | NK Cell Infusion
Number analyzed (Participants) | 21
participants
  Death | 1
  GvHD | 8

2. Secondary Outcome: Efficacy - Progression Free Survival
Description: Evaluate efficacy of natural killer (NK) cell infusions in terms of progression free survival (PFS) in number of months without disease progression.
Time Frame: 3 years
Population: Participants who completed cell infusion.
Measure: Mean (Full Range); unit: months
Arm/Group | NK Cell Infusion
Number analyzed (Participants) | 21
months | 12 [3 to 33]

3. Secondary Outcome: Efficacy - Overall Survival
Description: Evaluate efficacy of natural killer (NK) cell infusions in terms of overall survival (OS).
Time Frame: 8 years
Population: Participants who completed infusion. 9 patients were still alive at the time of this analysis.
Measure: Mean (Full Range); unit: months alive post-infusion
Arm/Group | NK Cell Infusion
Number analyzed (Participants) | 21
months alive post-infusion | 31 [2 to 92]

4. Secondary Outcome: Efficacy - Disease Progression
Description: Evaluate efficacy of natural killer (NK) cell infusions in terms of number of patients with disease progression.
Time Frame: 3 years
Population: Participants who completed cell infusion.
Measure: Number; unit: participants
Arm/Group | NK Cell Infusion
Number analyzed (Participants) | 21
participants | 10

ADVERSE EVENTS:
Time Frame: Each patient will be followed for toxicity until 8 weeks post-infusion or 5 months after the last natural killer cell infusion (NKI), whichever comes first. All adverse events will be recorded from the 1st day of infusion until the subject is off study.
Arm/Group | NK Cell Infusion
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cell Infusion (N=21)
Skin GVHD (Skin and subcutaneous tissue disorders) | 1 (1) — Acute Graft Versus Host Disease
Hemorrhage / Bleeding (Blood and lymphatic system disorders) | 1 (1)
Cardiac Left Ventricular Function (Cardiac disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NK Cell Infusion (N=21)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemolytic anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Infection - NOS (Infections and infestations) | 1 (1) — Mycobacterium in sputum culture
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 6 (7) — Parainfluenza; C-Diff; Varicella Zoster Virus; Cytomegalovirus; Gram negative bacteremia - Klebsiella
Infection - normal ANC - grade 1 or 2 neutrophils (Infections and infestations) | 5 (7) — Cytomegalovirus; Citrobacter; Fungal
Infection without Febrile Neutropenia (Infections and infestations) | 1 (1) — Polyoma Cystitis
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Acute Interstitial Nephritis (Metabolism and nutrition disorders) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Basal Cell Skin Cancer (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) — Fainting or Falling Down
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) — Hematuria
Protenuria (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) — Nocturia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes